CLINICAL TRIAL: NCT05379595
Title: A Phase 1b/2, Open-Label Study of Amivantamab Monotherapy and in Addition to Standard-of-Care Chemotherapy in Participants With Advanced or Metastatic Colorectal Cancer
Brief Title: A Study of Amivantamab Monotherapy and in Addition to Standard-of-Care Chemotherapy in Participants With Advanced or Metastatic Colorectal Cancer
Acronym: OrigAMI-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109215; 61186372GIC2002 (Other: Janssen Research & Development, LLC); 2021-006629-23 (EudraCT Number); 2023-506517-22-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2022-05-17; First posted 2022-05-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Advanced or Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — amivantamab; Fluorouracil; Leucovorin; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohorts A, B, and C: Amivantamab Monotherapy (Experimental): Participants with left-sided colorectal cancer (CRC) in Cohort A (no prior anti-epidermal growth factor receptor [EGFR] therapy) and in Cohort B (post anti-EGFR therapy), and right-sided CRC in Cohort C (with or without anti-EGFR therapy), will be administered intravenous (IV) infusion of amivantamab 1050 milligrams (mg) if body weight (BW) is less than (<) 80 kilograms (kg) or 1400 mg if BW is greater than or equal to (>=) 80 kg, as monotherapy on Days 1 and 15 of Cycle 2 (28-days cycle).
  Interventions: Biological: Amivantamab IV
- Cohorts Ph1b-D and D: Amivantamab+5-Fluorouracil, Leucovorin, and Oxaliplatin (mFOLFOX6) (Active Comparator): Participants who are anti-EGFR treatment naïve, have not received oxaliplatin-based chemotherapy in the metastatic setting, will be administered IV infusion of amivantamab 1050 or 700 mg (dose level 0 [DL0]) if BW is <80 kg, or 1400 or 1050 mg (dose de-escalation [DL-1]) if BW is >= 80 kg, on Days -1, -2, 8 and 22 of Cycle 1 and along with mFOLFOX6 SOC chemotherapy on Days 1 and 15 of Cycle 1 and Days 1 and 15 of Cycle 2 (each cycle of 28 days) in Phase 1b dose confirmation Cohort (Cohort Ph1b-D). Participant in Phase 2 Cohort (Cohort D) will receive recommended Phase 2 combination dose (RP2CD) of amivantamab along with mFOLFOX6 SOC chemotherapy determined in Cohort Ph1b-D.
  Interventions: Biological: Amivantamab IV; Biological: Fluorouracil; Biological: Leucovorin; Biological: Oxaliplatin
- Cohorts Ph1b-E and E: Amivantamab+5-Fluorouracil, Leucovorin, and Irinotecan (FOLFIRI) (Active Comparator): Participants who are anti-EGFR treatment naïve, have not received irinotecan-based chemotherapy in the metastatic setting, will be administered IV infusion of Amivantamab along with FOLFIRI SOC chemotherapy on Days -1, -2, and 8 of Cycle 1 and Days 1 and 15 of Cycle 2 in Ph1b-E. For Cohort E, RP2CD determined in Ph1b-E will be administered.
  Interventions: Biological: Amivantamab IV; Biological: Fluorouracil; Biological: Leucovorin; Biological: Irinotecan
- Cohort F: Amivantamab + mFOLFOX6 (Active Comparator): Participant who are treatment-naïve for right-sided unresectable or metastatic CRC. Participants will receive Amivantamab along with mFOLFOX6 SoC chemotherapy.
  Interventions: Biological: Fluorouracil; Biological: Leucovorin; Biological: Oxaliplatin; Biological: Amivantamab

INTERVENTIONS:
Biological: Amivantamab IV — Amivantamab will be administered as intravenous infusion.
  Other Names: RYBREVANT; JNJ-61186372
  Arms: Cohorts A, B, and C: Amivantamab Monotherapy; Cohorts Ph1b-D and D: Amivantamab+5-Fluorouracil, Leucovorin, and Oxaliplatin (mFOLFOX6); Cohorts Ph1b-E and E: Amivantamab+5-Fluorouracil, Leucovorin, and Irinotecan (FOLFIRI)
Biological: Fluorouracil — Fluorouracil will be administered as intravenous infusion.
  Arms: Cohort F: Amivantamab + mFOLFOX6; Cohorts Ph1b-D and D: Amivantamab+5-Fluorouracil, Leucovorin, and Oxaliplatin (mFOLFOX6); Cohorts Ph1b-E and E: Amivantamab+5-Fluorouracil, Leucovorin, and Irinotecan (FOLFIRI)
Biological: Leucovorin — Leucovorin will be administered as intravenous infusion.
  Arms: Cohort F: Amivantamab + mFOLFOX6; Cohorts Ph1b-D and D: Amivantamab+5-Fluorouracil, Leucovorin, and Oxaliplatin (mFOLFOX6); Cohorts Ph1b-E and E: Amivantamab+5-Fluorouracil, Leucovorin, and Irinotecan (FOLFIRI)
Biological: Oxaliplatin — Oxaliplatin will be administered as intravenous infusion.
  Arms: Cohort F: Amivantamab + mFOLFOX6; Cohorts Ph1b-D and D: Amivantamab+5-Fluorouracil, Leucovorin, and Oxaliplatin (mFOLFOX6)
Biological: Irinotecan — Irinotecan will be administered as intravenous infusion.
  Arms: Cohorts Ph1b-E and E: Amivantamab+5-Fluorouracil, Leucovorin, and Irinotecan (FOLFIRI)
Biological: Amivantamab — Amivantamab will be administered.
  Other Names: JNJ-61186372; RYBREVANT
  Arms: Cohort F: Amivantamab + mFOLFOX6

SUMMARY:
The purpose of this study is to assess the anti-tumor activity of amivantamab as a monotherapy (Cohorts A, B, and C), to assess the recommended phase 2 combination dose (RP2CD) of amivantamab when added to SoC chemotherapy (Ph1b cohorts) and to characterize the safety of amivantamab when added to standard-of care (SoC) chemotherapy in participants with metastatic colorectal cancer (mCRC) (Ph2 cohorts).

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is a major global health concern and the third most common cancer worldwide. Amivantamab (also known as RYBREVANT or JNJ-61186372) is a fully human immunoglobulin (Ig) G1-based bispecific antibody (Ab) directed against the epidermal growth factor (EGF) and mesenchymal epithelial transition (MET) receptors, with evidence of preclinical activity against non-small cell lung cancer (NSCLC) tumors with activating EGF receptor (EGFR) mutations, the T790M and C797S second-site resistance EGFR mutations, overexpressed wild-type EGFR, as well as with activation of the MET pathway. Amivantamab has demonstrated activity in both EGFR- and MET-driven NSCLC, with preclinical evidence demonstrating its ability to recruit immune effector cells. While two anti-EGFR antibodies are incorporated as part of the SoC for CRC patients, MET is highly expressed or amplified in subsets of CRC and additionally plays a role in mediating resistance to anti-EGFR treatments. The study consists of up to 28 days screening period, treatment period will begin on Cycle 1 Day 1 (C1D1) (for Cohorts A, B, and C) or C1D -2 (for Ph1b-D, Ph1b-E, Cohorts D, E and F) with the administration of the study treatment and continue as 28-day cycles until the end of treatment visit, up to 30 days after discontinuation of study treatment. The safety of amivantamab as a monotherapy or in addition to SoC chemotherapy will be assessed by physical examinations, Eastern Cooperative Oncology Group (ECOG) criteria for performance status (PS), laboratory tests, vital signs, monitoring of adverse events, and concomitant medication usage.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have been previously diagnosed with histologically or cytologically confirmed unresectable or metastatic adenocarcinoma of the colon or rectum
* Participant must have tumor previously characterized as having wild-type Kirsten rat sarcoma viral oncogene (KRAS), neuroblastoma RAS viral oncogene homolog (NRAS), v-raf murine sarcoma viral oncogene homolog B (BRAF), and without evidence of Erb-b2 receptor tyrosine kinase 2/human epidermal growth factor receptor 2 (ERBB2/HER2) amplification. Additional cohort-specific requirements:

  * Phase (Ph) 2 (Cohorts A, B, and C) Amivantamab monotherapy: Participant must have received at least 2 but not more than 3 prior lines of systemic therapy in the metastatic setting. Participant must have been diagnosed with left-sided colorectal cancer (CRC) (Cohort A and B) and right-sided (Cohort C)and have received or been intolerant to standard of care (SoC) fluoropyrimidine-, oxaliplatin-, and irinotecan-based chemotherapy and an anti-vascular endothelial growth factor (VEGF) treatment. Participant must be anti-EGFR treatment naive in Cohort A, an anti-epidermal growth factor receptor (EGFR) treatment Cohort B, with or without an anti-EGFR treatment in Cohort C
  * Ph 1b Dose Confirmation Cohorts (Ph1b-D and Ph1b-E), Ph2 (Cohorts D and E) Amivantamab+mFOLFOX6/FOLFIRI: Participant must been diagnosed with CRC and have received no more than 1 prior line of systemic therapy in the metastatic setting. Cohort Ph1b-D/Cohort D: Participant must be anti-EGFR treatment naïve, have not received oxaliplatin-based chemotherapy in the metastatic setting, and be eligible for treatment with mFOLFOX6 according to local regulatory approvals and SoC guidelines. Cohort Ph1b-E/Cohort E: Participant must be anti-EGFR treatment naïve, have not received irinotecan-based chemotherapy in the metastatic setting, and be eligible for treatment with FOLFIRI according to local regulatory approvals and SoC guidelines
  * Ph2 Cohorts F Amivantamab subcutaneous (SC) + mFOLFOX6: Participants must be treatment-naive for right-sided unresectable or metastatic CRC and be eligible for treatment with mFOLFOX6 according to local regulatory approvals and SoC guidelines
* For Phase 1 dose confirmation cohorts (Cohorts Ph1b-D and Ph1b-E): Participant must have evaluable disease. For Phase 2: Participant must have measurable disease according to Response Criteria in Solid Tumors (RECIST) Version 1.1. If only one measurable lesion exists, it may be used for the screening biopsy as long as baseline tumor assessment scans are performed greater than or equal to (>=) 7 days after the biopsy
* Participant must have Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Participant must have a tumor lesion amenable for biopsy and agree to mandatory protocol-defined screening biopsy. Biopsies are required if clinically feasible for participants in Ph1b-D, Ph1b-E, and Cohort F. For Cohort F, archival tissue is required if a fresh biopsy is not feasible
* A female participant of childbearing potential must have a negative serum pregnancy test at screening and within 72 hours of the first dose of study treatment and must agree to further serum or urine pregnancy tests during the study. Note: Participant must not be pregnant, breastfeeding, or planning to become pregnant while enrolled in this study

Exclusion Criteria:

* Cohorts A, B, C, Ph1b-D, D, Ph1b-E, and E: Participant with identified mutation in Kirsten rat sarcoma viral oncogene (KRAS), neuroblastoma RAS viral oncogene homolog (NRAS), v-raf murine sarcoma viral oncogene homolog B (BRAF), or epidermal growth factor receptor (EGFR) ectodomain, or ERBB2/HER2 amplification by central circulating tumor deoxyribonucleic acid (ctDNA) testing at screening; Cohort F: Participant with identified mutation in KRAS, NRAS, BRAF V600, or PTEN, identified fusions in ALK, ROS-1, RET, and NTRK 1, ERBB2/HER2 amplification, or identified to have MSI-H status by central ctDNA testing at screening
* Participant with symptomatic or untreated brain metastasis
* History or known presence of leptomeningeal disease
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (for example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2027-04-27 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Cohorts A, B, and C: Objective Response Rate (ORR) | Up to 4 years 3 months
  ORR is defined as the percentage of participants who achieve either a partial response (PR) or complete response (CR), as defined by investigator assessment using Response Criteria in Solid Tumors (RECIST) version 1.1.
Cohorts Ph1b-D and Ph1b-E: Number of Participants with Dose-limiting Toxicity (DLT) | Up to 4 years 3 months
  Number of participants with DLT will be assessed. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.
Cohorts Ph1b-D and Ph1b-E: Number of Participants with DLT by Severity | Up to 4 years 3 months
  Number of participants with DLT by severity will be assessed. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity. Toxicities will be graded for severity according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0, graded as Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: life-threatening, and Grade 5: death related to adverse event.
Cohorts D and E: Number of Participants with Adverse Events (AE) | Up to 4 years 3 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study. Severity of AEs will be graded according to the NCI CTCAE version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: life-threatening and Grade 5: death related to adverse event.
Cohorts D and E: Number of Participants with Laboratory Values Abnormalities | Up to 4 years 3 months
  Number of participants with laboratory values abnormalities, which includes serum chemistry, hematology, coagulation, and urinalysis, will be reported.
Cohorts D and E: Number of Participants with Vital Signs Abnormalities | Up to 4 years 3 months
  Number of participants with vital signs including temperature, heart rate, respiratory rate, and blood pressure (systolic and diastolic) and oxygen saturation, abnormalities will be reported.
Cohorts F: Number of Participants with Adverse Events (AE) | Up to 4 years 3 months
  An AE is any untoward medical occurrence in a participant taking part in a in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study. Severity of AEs will be graded according to the NCI-CTCAE version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: life-threatening and Grade 5: death related to adverse event.
Cohorts F: Number of Participants with Laboratory Values Abnormalities | Up to 4 years 3 months
  Number of participants with laboratory values abnormalities, which includes serum chemistry, hematology, coagulation, and urinalysis, will be reported.
Cohorts F: Number of Participants with Vital Signs Abnormalities | Up to 4 years 3 months
  Number of participants with vital signs including temperature, heart rate, respiratory rate, and blood pressure (systolic and diastolic) and oxygen saturation, abnormalities will be reported.

SECONDARY OUTCOMES:
Cohorts A, B, C, Ph1b-D, and Ph1b-E: Number of Participants with AEs | Up to 4 years 3 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study. Severity of AEs will be graded according to the NCI CTCAE version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: life-threatening and Grade 5: death related to adverse event.
Cohorts A, B, C, Ph1b-D, and Ph1b-E: Number of Participants with Laboratory Values Abnormalities | Up to 4 years 3 months
  Number of participants with laboratory values abnormalities, which includes serum chemistry, hematology, coagulation, and urinalysis, will be reported.
Cohorts A, B, C, Ph1b-D, and Ph1b-E: Number of Participants with Vital Signs Abnormalities | Up to 4 years 3 months
  Number of participants with vital signs including temperature, heart rate, respiratory rate, and blood pressure (systolic and diastolic) and oxygen saturation, abnormalities will be reported.
Cohorts Ph1b-D, Ph1b-E, D, E and F: ORR | Up to 4 years 3 months
  ORR is defined as the percentage of participants who achieve either a PR or CR, as defined by investigator assessment using RECIST version 1.1.
Cohorts Ph1b-D, Ph1b-E, D, E and F: Duration of Response (DoR) | Up to 4 years 3 months
  DoR is defined as the time from the date of first documented response (PR or CR) until the date of documented progression or death, whichever comes first, for participants who have PR or CR, as defined by investigator assessment using RECIST version 1.1.
Cohorts Ph1b-D, Ph1b-E, D, E and F: Disease Control Rate (DCR) | Up to 4 years 3 months
  DCR is defined as the percentage of participants achieving a best overall response (BOR) of CR, PR or stable disease (with minimum duration of 7 weeks) as defined by RECIST v1.1.
Cohorts Ph1b-D, Ph1b-E, D, E and F: Clinical Benefit Rate (CBR) | Up to 4 years 3 months
  CBR is defined as the percentage of participants achieving complete or partial response, as well as durable stable disease (defined as a duration of at least 11 weeks) as defined by RECIST version 1.1.
Cohorts D, E and F: Progression Free Survival (PFS) | Up to 4 years 3 months
  PFS is defined as the time from the first administration of study treatment until the date of objective disease progression or death, whichever comes first, based on investigator assessment using RECIST version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (53):
- United States (14):
  - O Neal Comprehensive Cancer Center at UAB, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles UCLA, Los Angeles, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - University of Maryland School of Medicine, Baltimore, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - Start Midwest, Grand Rapids, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - NYU Langone Long Island Clinical Research Associates, New York, New York
  - Herbert Irving Comprehensive Cancer Center Columbia University Medical Center, New York, New York
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Belgium (4):
  - Institut Jules Bordet, Anderlecht
  - Cliniques Universitaires Saint Luc, Brussels
  - UZ Antwerpen, Edegem
  - Universitair Ziekenhuis Gasthuisberg, Leuven
- Canada (3):
  - BC Cancer Agency - Vancouver BC, Vancouver, British Columbia
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre University Health Network, Toronto, Ontario
- China (4):
  - The Second Hospital To Dalian Medical University, Dalian
  - Sun Yat-sen University - The Sixth Affiliated Hospital Guangdong Gastrointestinal Hospital, Guangzhou
  - The Second Affiliated Hospital of Zhejiang University College of Medicine, Hangzhou
  - Hubei province tumor hospital, Wuhan
- Germany (2):
  - Asklepios Klinik Altona, Hamburg
  - Ludwig-Maximilians-Universitaet Muenchen, Munich
- Italy (3):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - A O Ospedale Niguarda Ca Granda, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
- Malaysia (3):
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Umum Sarawak, Kuching
  - Beacon Hospital Sdn Bhd, Petaling Jaya
- Puerto Rico (2):
  - Ad Vance Medical Research, Ponce
  - Pan American Center for Oncology Trials LLC, Rio Piedras
- South Korea (5):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
- Spain (7):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp Univ Hm Sanchinarro, Madrid
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Clinico Univ. de Valencia, Valencia
- Taiwan (6):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chi Mei Medical Center Liu Ying, Liou Ying Township
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency